CLINICAL TRIAL: NCT02531711
Title: Chronic Lumbosacral Radiculopathy: Impact of an Analgesic Dietary Intervention on Pain & Function
Acronym: LRPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: North American Spine Society (NASS) (Unknown); Mayday Fund (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 14-2321
Record Dates: First submitted 2015-06-08; First posted 2015-08-24 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Pain
Keywords: Lumbosacral; radicular
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diet A (Experimental): Dietary intervention: Dietary fats are adjusted. Key study foods and oils are provided for 12 weeks. Participants learn which foods to eat and which to avoid.
  Interventions: Other: Diet A
- Diet B (Active Comparator): Dietary intervention: This diet also adjusts dietary fats, and provides key study foods and oils for 12 weeks.
  Interventions: Other: Diet B

INTERVENTIONS:
Other: Diet A — Experimental analgesic dietary intervention
  Arms: Diet A
Other: Diet B — Healthy comparator diet
  Arms: Diet B

SUMMARY:
The goal of this proposed research is to assess the preliminary efficacy of dietary interventions that change dietary fats in improving clinical outcomes related to lumbar radicular pain. After a two-week baseline, consented participants are randomized to one of two diets. Key foods consistent with the diet are provided for 12 weeks along with extensive dietary counseling and support from the study-provided materials. Participants are encouraged to follow the assigned diet for another 6 weeks without provision of food.

Participants complete questionnaires at baseline, randomization, and after 6 weeks, 12 weeks, and 18 weeks on the diet. They provide blood samples at randomization (2 weeks) and after 12 and 18 weeks on the diet.

DETAILED DESCRIPTION:
Lumbar radiculopathy is a fairly common pain syndrome which may result in chronic, severe disability. There are few successful treatment options for patients with persistent lumbosacral radicular pain (LRP) that does not respond to conventional approaches. A fundamental biologic mechanism of chronic LRP, as well as other chronic pain syndromes, may involve failure of inflammation-resolution, an active process driven by lipid mediators derived from fatty acids (resolvins, protectins, maresins). The investigators' preliminary studies indicate that dietary modifications, specifically increasing some dietary fatty acids, while reducing others, result in large, statistically significant and clinically relevant improvement in headache frequency, intensity, and other clinical outcomes in community dwelling persons with chronic headaches.

The proposed trial represents a promising approach to treatment of a disabling condition, lumbar radiculopathy. The previous headache trial by the investigators' interdisciplinary UNC/NIH team demonstrated that specific dietary manipulations can produce marked biochemical changes and have a major positive clinical impact. This project promises to enhance the generalizability of the investigators' approach by expanding from chronic headaches to another common chronic pain condition, and also by using a more cost-effective intervention. Because dietary modification is a relatively safe and low-cost health-improvement strategy, the long-term outcome of this research may be to empower individuals to take a more active role in their own health through dietary changes that reduce dependence on medical treatments, while providing significant clinical benefits.

Baseline Phase. Medical records will be obtained for the participant's history and physical examination (performed by referring physician at the Spine Center). The baseline visit will consist of review of inclusion/exclusion criteria and the components of the study prior to consenting. Those who wish to sign the consents will complete baseline assessment instruments that measure lumbosacral radiculopathy characteristics and their impact on quality-of-life. Through electronic diaries, participants will provide daily data on pain intensity, duration, function, sleep quality, and medication use over a 2-week baseline phase. Participants who are compliant with all aspects of data collection, and who experience daily radicular pain, will be eligible for study intervention participation.

Randomization. At the end of the 2-week baseline phase, participants who qualify will be randomized (computer-generated variable permuted block) to: 1) the High n-3, Low n-6 Diet (Analgesic Diet); or 2) the Control Diet. Blood will be collected for baseline biomarker assessment prior to beginning study diets.

Post Randomization. After randomization, participants will attend an initial, in-depth dietary counseling session administered by the registered dietitian. Participants will be asked to provide a dietary history and will receive detailed instruction in the specific dietary intervention per group assignment. Participants in each group will attend a total of 3 in-person follow-up sessions with the dietitian, for review of their dietary experiences, to receive encouragement, to clarify issues, and to have questions answered. At each visit, the dietitian will obtain a dietary history and assessment, provide tailored counseling, and record data for evaluation of participant variability in order to guide future sessions. Participants will have a visit with the dietitian at randomization, two weeks later, 4 weeks after that, and 6 weeks after that (at the end of the intervention). In addition, individuals will participate in brief (15-20 minute) check-in telephone calls with the dietitian every 2-3 weeks. Participants will have contact with the research assistant twice weekly to encourage diary completion and to invite adverse event reporting.

During the 12-week intervention phase (weeks 2-14), participants will be provided with essential foods to enable them to follow diet recommendations, including study oils, salad dressings, and unprepared protein sources (meat, beans, fish). For the remainder of their meals, participants will choose food products consistent with their assigned diet. At the conclusion of the post-intervention phase (Week 20, Diet week 18), participants will complete on-line questionnaires and provide blood samples. The purpose of this post-intervention phase is: 1) to obtain pilot data on the ability of participants to continue to achieve nutrient intake targets without counseling and food provision; and 2) to obtain pilot data on the post-intervention trajectory of biochemical and clinical outcomes.

Throughout the 12-week active intervention and the 6-week post-intervention phases, participants will have access to detailed intervention materials. Diet education materials include the diet guidelines, allowed food list, how to read food labels, grocery shopping guides for 9 local grocery stores, dining out guide, 7-day meal plan and 75 recipes with the ability for the dietitian to add more.

Food Supply. Participants will visit the dietitian 3 times during the 12-week active intervention to obtain specific food items with targeted nutrient compositions. Food items will include: cooking oils, salad dressings, mayonnaise, portable dressing packets, unprepared frozen food items, and key ingredients for home preparation of meals and snacks. All foods have been specifically selected to ensure that participants meet specific nutrient intake targets. Prior nutrient analyses of more than 80 relevant food items was performed as part of the investigators' previous dietary intervention study in participants with chronic daily headache, by the National Institutes of Health-National Institute on Alcohol Abuse and Alcoholism Section of Nutritional Neurosciences (SNN). The SNN has agreed to provide further nutrient analysis as needed for the proposed study.

Assessments. Throughout the 2-week baseline, the 12-week active intervention, and 6-week post-intervention phases, all participants will record pain intensity, pain interference, medication use, activity, and stress using a daily pain diary accessed by mobile device.

Blood samples will be collected during three visits at the end of the baseline phase (Week 2, Diet week 0) and then at study Weeks 14 and 20 (at the end of the active intervention and at the end of the post-intervention period) for nutritional and metabolic biomarker measurement. At each sample collection visit (and after 6 weeks on the diet), participants will also complete the Oswestry Disability Index (ODI) and NIH PROMIS-29 battery (physical function, anxiety, depression, fatigue, sleep disturbance, satisfaction with social role, pain interference, pain intensity). Every 6 weeks, participants will also be asked about their use of other modalities for pain control, including physical therapy, spinal manipulation, epidural corticosteroid injections, acupuncture, and yoga.

Interventions. All participants will receive: 1) tailored dietitian-administered counseling consistent with the group assignment; 2) access to intervention-specific informational materials and daily outcome assessments; and 3) critical food items with precisely quantified fatty acid composition, selected to meet nutrient intake targets specific for each of the assignment groups.

Random Allocation. At the first intervention visit, At Week 2, the research dietitian will enter the participant's assigned ID into an online computer program that will determine assignment to one of the two diets. Using a random number sequence to generate a permuted block of 2-4, the program ensures equal numbers of participants in each arm. The program documents treatment assignment in an un-editable form including a date stamp.

Masking. The research staff, masked to treatment assignment, will schedule all study-related visits in the Clinical and Translational Research Center (CTRC) or other appropriate site in the University of North Carolina (UNC) Healthcare system or medical school. Only the dietitian will, of necessity, be unmasked. All investigators and laboratory personnel will be masked to dietary assignment. Masking will be maintained in the random allocation procedure. The research dietitian will not indicate to participants which diets are considered to be treatment diets vs. the control diet.

ELIGIBILITY:
Inclusion Criteria:

MRI-verified lumbosacral radiculopathy associated with herniated disc, spinal stenosis, or post-surgical fibrosis

* Pain reaching to the knee for at least 12 weeks
* Willing to complete daily diary for 20 weeks, as evidenced by completion of ≥12 of the first 14 days
* Possessing a mobile device (smart phone, tablet, laptop) capable of accessing the application and website
* Able to attend dietitian counseling sessions in Chapel Hill, NC
* Under care of a physician for LR
* Able to read and communicate in English

Exclusion Criteria:

* Psychosis or severe depression, anxiety, substance abuse disorder
* History of specific food allergies that would prevent adherence to study diet
* Aversion to eating fish
* Currently taking fish oil or other supplements that contain fatty acids under investigation
* Pregnancy or anticipated pregnancy
* Active treatment for a major medical illness, such as malignancy, autoimmune, immune deficiency disorder
* History of vasculitis, intracranial mass, clotting disorder (including medication-induced, e.g., warfarin)
* Cognitive dysfunction preventing informed consent
* Pending personal injury litigation, including worker's compensation
* Chronic long-term disability related to lumbosacral injury/symptoms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Oswestry Disability Index--Primary clinical outcome | 12 weeks
  Measure of pain-specific quality of life
17-Hydroxy Docosahexaenoic acid (DHA)--Primary biochemical outcome | 12 weeks
  Metabolite related to dietary fatty acid intakes implicated in pain reductions

SECONDARY OUTCOMES:
Pain intensity | 12 weeks
  Average weekly pain intensity, measured in daily diary
Physical activity | 12 weeks
  Average weekly steps per day, measured by pedometer (Fitbit)
Sleep efficiency | 12 weeks
  Measured by percent of time asleep out of total time in bed (Fitbit)
Sleep quantity | 12 weeks
  Measured by average weekly hours of sleep (Fitbit)
Self-reported health | 12 weeks
  PROMIS-29: includes physical function, social functioning, psychological distress, sleep quality, and fatigue
Red blood cell fatty acids | Measured at Week 2 and after 6 and 12 weeks on the diet
  Measures adherence to dietary recommendations
Borkovec and Nau scale | Measured at Week 2
  Measures credibility and expectation of benefit

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Carneiro, DO, Principal Investigator — Department of Physical Medicine and Rehabilitation, University of North Carolina at Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be shared with investigators at NIH.